CLINICAL TRIAL: NCT01808664
Title: Promoting Patient-Centered Counseling to Reduce Inappropriate Diagnostic Tests: Randomized Clinical Trial
Brief Title: Promoting Patient-Centered Counseling to Reduce Inappropriate Diagnostic Tests
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Davis (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Health Services Research
Other Study IDs: 364498; 364498-3 (Other: UC Davis)
Record Dates: First submitted 2012-11-20; First posted 2013-03-11 (Estimated); Last update posted 2020-02-26 (Actual); Status verified 2020-02

CONDITIONS: Unnecessary Procedures; Low Back Pain; Osteoporosis; Headache; Magnetic Resonance Imaging; Primary Care
MeSH Terms: conditions — Low Back Pain; Osteoporosis; Headache

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Standardized Patient Instructor Intervention (Experimental): Primary care physicians (PCPs) randomized to intervention will receive over a three month run-in period two visits by standardized patient instructors portraying: 1) a 48 year-old patient with low back pain for less than six-weeks and no "red flags" for immediate spinal imaging; and 2) a 50 year-old recently menopausal woman establishing care with concerns about osteoporosis risk.
  Interventions: Behavioral: Standardized Patient Instructor Intervention
- Control (Active Comparator): In the latter half of visits with control PCPs, standardized patient instructors (SPIs) will share information regarding low back pain or bone health that are unrelated to diagnostic testing, but will not discuss patient-centered techniques or conduct training. The total duration of the control "information sharing" will be about one-third the SPI intervention to enhance patient-centeredness.
  Interventions: Behavioral: Control

INTERVENTIONS:
Behavioral: Standardized Patient Instructor Intervention — In each case, patients will harbor underlying concerns about a serious underlying condition (e.g., either disc herniation or osteoporosis) and will request inappropriate tests. Standardized patient instructors (SPIs) will portray new patients visiting the clinic for the first time, and electronic medical records will be identical to that of actual new patients.
  During the initial part of intervention visits, SPIs will assess the extent to which PCPs engage in patient-centered techniques specified in the final intervention model. SPIs will then break of their role and either teach or reinforce PCP use of the techniques, presenting techniques in a logical sequence while emphasizing flexibility in their use. SPIs will use scripts to deliver the interventions, providing opportunities for PCPs to ask questions, discuss concepts, and practice (by role playing) patient-centered techniques.
  Arms: Standardized Patient Instructor Intervention
Behavioral: Control — In the latter half of visits with control PCPs, standardized patient instructors will share information with physicians regarding the acute low back pain self-care and bone health, but will not discuss patient-centered techniques or conduct training. The total duration of the control "information sharing" will be about one-third the SPI intervention to enhance patient-centeredness.
  Arms: Control

SUMMARY:
In this study, the investigators will develop and evaluate a novel intervention using standardized patients (SPs) -- or actors playing the roles of patients -- to enhance physicians' patient-centered counseling skills regarding two frequently overused, potentially inappropriate services in primary care: magnetic resonance imaging (MRI) for acute low back pain and bone densitometry in women at low-risk for osteoporosis. The investigators will further evaluate whether intervention effects on physician patient-centeredness generalize to counseling regarding other costly, unnecessary diagnostic tests.

ELIGIBILITY:
Inclusion Criteria:

* Resident physician in family medicine or internal medicine who deliver primary care at one of two hospital-based primary care clinics at the University of California, Davis Medical Center Sacramento

Exclusion Criteria:

* Anticipated graduation in less than one year from enrollment.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2013-04; Primary Completion 2014-09 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Number of inappropriate diagnostic tests ordered | 9 months
  Investigators will assess via blinded, standardized chart review whether study physicians ordered inappropriate diagnostic tests for unannounced standardized patients who request testing during three follow-up visits occurring 3 to 9 months post-randomization.

SECONDARY OUTCOMES:
Use of patient-centered counseling techniques | 9 months
  Physician use of patient-centered counseling techniques as assessed via masked recordings of three standardized patient visits
Actual diagnostic test ordering among real patients | 9 months post-intervention
  Among real patients seen by study physicians, we will assess diagnostic test ordering among actual adult patients during the post-intervention period. We will also assess comparable diagnostic test ordering during the pre-intervention period to enable adjustment for baseline test ordering.

OTHER OUTCOMES:
Standardized Patient Satisfaction | 9 months
  Standardized patients will complete a measure of patient satisfaction based on the Consumer Assessment of Health Plans Survey (CAHPS) during each of three unannounced visits occuring during the follow-up period

CONTACTS AND LOCATIONS:
Overall Officials: Joshua J Fenton, MD, MPH, Principal Investigator — University of California, Davis

REFERENCES:
- [Background] May L, Franks P, Jerant A, Fenton J. Watchful Waiting Strategy May Reduce Low-Value Diagnostic Testing. J Am Board Fam Med. 2016 Nov 12;29(6):710-717. doi: 10.3122/jabfm.2016.06.160056. PMID 28076254
- [Result] Fenton JJ, Kravitz RL, Jerant A, Paterniti DA, Bang H, Williams D, Epstein RM, Franks P. Promoting Patient-Centered Counseling to Reduce Use of Low-Value Diagnostic Tests: A Randomized Clinical Trial. JAMA Intern Med. 2016 Feb;176(2):191-7. doi: 10.1001/jamainternmed.2015.6840. PMID 26640973